CLINICAL TRIAL: NCT01665846
Title: Neuroimaging Correlates of Monocyte/Macrophage Infiltration in HIV-infected Individuals: A Cross-sectional Pilot Study Using IV Ferumoxytol
Brief Title: Ferumoxytol-enhanced Brain MRI in HIV-associated Neurocognitive Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Beau Nakamoto, Assistant Professor, University of Hawaii
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H015
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: HIV Dementia
Keywords: HIV associated neurocognitive disorders; MRI; Ferumoxytol
MeSH Terms: conditions — AIDS Dementia Complex | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ferumoxotyol (Experimental): Brain MRI will be performed before and 48 +/- 8 hours after ferumoxytol administration.
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol — A dose of 4 mg/kg of ferumoxytol up to a maximum of 510 mg of elemental iron will be administered.
  Other Names: FERAHEME

SUMMARY:
The purpose of this study is to describe the radiologic findings on brain MRI after ferumoxytol administration in HIV-infected patients with cognitive impairment.

DETAILED DESCRIPTION:
The continued existence of cognitive dysfunction in HIV infected individuals in the era of effective antiretroviral therapy may be, in part, secondary to the failure of current antiretroviral regimens to eradicate the pool of HIV-infected and activated monocytes within the bloodstream. Trafficking of such HIV infected and activated blood monocytes into the brain parenchyma is believed to introduce HIV into the brain and precipitate immune activation and inflammation, ultimately leading to neuronal degeneration.

Ferumoxytol is an ultrasmall superparamagnetic iron-oxide (USPIO), which is FDA-approved for intravenous iron-replacement therapy in anemic patients with chronic kidney disease. The paramagnetic properties of ferumoxytol also allow it to be used as a MRI contrast agent. Ferumoxytol is avidly taken up by circulating monocytes and reactive astrocytes, microglia, and dendritic cells within the brain, making it potentially a novel biomarker for HIV-associated cognitive impairment given the role of monocytes in its pathogenesis.

This proposal intends to investigate the possible use of ferumoxytol (a new MRI contrast agent) as a biomarker for HIV-associated cognitive impairment and to assess the safety and tolerability of ferumoxytol in HIV-infected individuals.

Hypotheses to be tested:

* HIV-infected subjects with undetectable plasma HIV RNA levels and detectable levels of HIV DNA in CD14+ peripheral blood mononuclear cells (PBMCs) and impairment on neurocognitive testing will demonstrate ferumoxytol contrast enhancement in the perivascular regions of the brain consistent with monocyte/macrophage infiltration in these regions.
* Ferumoxytol can be safely administered to HIV-infected subjects.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection as documented by ELISA and confirmed by Western blot, HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA by RT-PCR or DNA at any time prior to study entry.
* Receipt of antiretroviral (ARV) medication uninterrupted for at least 6 months leading up to the screening period with demonstrated plasma HIV RNA < 48 copies/ml within the last 6 months.
* Willingness for both males and females of childbearing potential to utilize 2 effective contraception methods (2 separate forms, one of which must be an effective barrier method), be non-heterosexually active or have a an exclusive vasectomized partner from screening throughout the duration of the study treatment and for 30 days following the last dose of study drugs.
* Age >18 years.
* Ability and willingness to provide written informed consent
* HIV DNA > 10 copies/106 CD14+ PBMCs
* Mild or greater cognitive impairment as indicated by global NPZ8 z-score < -0.5 with a neurocognitive abnormality (defined as a z-score < -0.5) in at least one cognitive domain characteristic of HAD (i.e., executive function, psychomotor speed, memory).

Exclusion Criteria:

* Requirement for acute therapy for other AIDS-defining illness or other serious medical illnesses (in the opinion of the site investigator) within 14 days prior to study entry.
* Known allergic or hypersensitivity reaction to FERAHEME, parental iron, parental dextran, parental iron-dextran, or parental iron-polysaccharide preparations
* Known history of an iron overload syndrome (e.g., hereditary hemochromatosis, porphyria cutanea tarda)
* Medical conditions (e.g., chronic hemolytic anemia) which requires frequent blood transfusions
* Taking oral iron supplementation
* Any factor that precludes MRI scan including presence of metal or exposure to metal work (e.g. metal grinder/worker) and claustrophobia
* Past or present HIV opportunistic infection of the brain, learning disability, head injury with prolonged loss of consciousness or cognitive sequelae, or other non-HIV risk factor that in the opinion of the principal investigator (PI) may impact cognitive performance.
* History of epilepsy requiring treatment with an antiepileptic
* Other chronic illnesses including insulin-dependent diabetes, autoimmune diseases, and endocrinopathies, except subjects on stable physiologic replacement therapy for low testosterone or thyroid levels
* Current active substance or alcohol dependence or positive urine toxicology screen.
* Pregnancy or breast-feeding, intent to become pregnant during the course of the study.
* Any condition which, in the opinion of the investigator, would compromise the subject's ability to participate in the study
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) greater than 2x upper limits of normal on pre-entry baseline laboratory safety assessment prior to study enrollment.
* Elevated iron levels on pre-entry baseline laboratory safety assessment prior to study enrollment.
* Hematocrit > 52% or Hemoglobin > 18 g/dL on pre-entry baseline laboratory safety assessment prior to study enrollment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Post-ferumoxytol enhancement on Brain MRI | 48 hour following administration of a dose of 4 mg/kg of feruomoxytol up to a maximum of 510 mg of elemental iron
  The location and extent of ferumoxytol enhancement within the brain will be described.

SECONDARY OUTCOMES:
Safety | 1 hour and 1 month following administration of a dose of 4 mg/kg of ferumxotyol up to a maximum of 510 mg of elemental iron
  The rate of overall grade > 2 toxicities (categorized by the NIAID Division of AIDS adverse events table) during ferumoxytol infusion and 1 month post-ferumoxytol infusion will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Beau K Nakamoto, MD, PhD, Principal Investigator — University of Hawaii, Hawaii Center for AIDS, John A Burns School of Medicine
Locations (1):
- Hawaii Center for AIDS, Honolulu, Hawaii, United States

REFERENCES:
- [Background] Neuwelt EA, Hamilton BE, Varallyay CG, Rooney WR, Edelman RD, Jacobs PM, Watnick SG. Ultrasmall superparamagnetic iron oxides (USPIOs): a future alternative magnetic resonance (MR) contrast agent for patients at risk for nephrogenic systemic fibrosis (NSF)? Kidney Int. 2009 Mar;75(5):465-74. doi: 10.1038/ki.2008.496. Epub 2008 Oct 8. PMID 18843256
- See also: AMAG Pharmaceuticals — http://www.amagpharma.com/products/ferumoxytol.php